CLINICAL TRIAL: NCT03417505
Title: Tangible Hydra-PEG: A Promising Solution for Scleral Lens Wearers With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tangible Science (Industry)
Collaborators: Nova Southeastern University (Other); University of California, Davis (Other); Illinois College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: STM-0686
Record Dates: First submitted 2018-01-10; First posted 2018-01-31 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye; Dry Eye Syndromes
Keywords: Contact lens discomfort; Scleral lens; Tangible Hydra-PEG
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked crossover study
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treated followed by untreated (Experimental): Patients wear the Hydra-PEG treated scleral lenses for 30 days. After testing and a post contact lens wear washout period, these patients will then wear the untreated lenses for 30 days. In this arm, the intervention (scleral lenses treated with Tangible Hydra-PEG) is administered prior to the control treatment (untreated scleral lenses).
  Interventions: Device: Scleral lenses treated with Tangible Hydra-PEG; Device: Untreated scleral lenses
- Untreated followed by treated (Experimental): Patients wear the untreated scleral lenses for 30 days. After testing and a post contact lens wear washout period, these patients will then wear the Hydra-PEG treated lenses for 30 days. In this arm, the intervention (scleral lenses treated with Tangible Hydra-PEG) is administered after the control treatment (untreated scleral lenses).
  Interventions: Device: Scleral lenses treated with Tangible Hydra-PEG; Device: Untreated scleral lenses

INTERVENTIONS:
Device: Scleral lenses treated with Tangible Hydra-PEG — Scleral lenses treated with Tangible Hydra-PEG, a hydrophilic, PEG-based contact lens coating designed to improve lens wettability, deposit resistance, and tear film breakup time.
  Other Names: Tangible Hydra-PEG is a hydrophilic PEG-based lens coating
Device: Untreated scleral lenses — Scleral lenses without the Tangible Hydra-PEG treatment will serve as a control.
  Other Names: control

SUMMARY:
Tangible Hydra-PEG is a novel coating technology designed to improve lens wettability, deposit resistance, and tear film breakup time. This is a randomized double masked cross-over study to examine contact lens discomfort and dry eye symptoms with Tangible Hydra-PEG treated scleral lens wear compared to untreated scleral lens wear in the dry eye patient population.

DETAILED DESCRIPTION:
Dry eye (DE) is a common complaint of millions of people worldwide with a significant impact on quality of life. For decades, this condition has presented a challenge to eye care professionals as conventional therapies are often ineffective. Recently, scleral lenses have demonstrated to be a promising therapeutic and vision rehabilitative option for dry eye sufferers. Nonetheless, despite the benefits of scleral lenses for dry eye patients, inadequate wettability of scleral lenses with subsequent diminished comfort and visual clarity remains a concern for scleral lens wearers with dry eye.

Tangible Hydra-PEG (Tangible Science LLC, Menlo Park, CA, USA) is a novel coating technology designed to improve lens wettability, deposit resistance, and tear film breakup time, ultimately enhancing contact lens comfort. While studies have shown that Tangible Hydra-PEG technology can improve contact lens discomfort (CLD) in soft contact lens and gas permeable lens wearers, to our knowledge, no clinical research investigation has examined the benefits of this new coating on scleral lens wear in dry eye sufferers. As such, the aim of this study is to compare the CLD and DE symptoms of dry eye scleral lens wearers between Tangible Hydra-PEG treated scleral lens wear and untreated scleral lens wear. CLD and DE signs will also be assessed to corroborate our findings.

This will be the first randomized double masked cross-over study to examine CLD and DE symptoms of Tangible Hydra-PEG treated scleral lens wear compared to untreated scleral lens wear in the dry eye patient population. Tangible Hydra-PEG treated scleral lenses can potentially minimize CLD and DE symptoms, ultimately improving outcomes for patients coping with dry eye disease. This study will provide new information about this innovative technology and help practitioners envisage rehabilitative options which will best optimize the quality of life of this important patient population.

ELIGIBILITY:
Inclusion Criteria:

* Reduced tear film break up time (TBUT), a sign of dry eye disease and contact lens discomfort
* Scleral lens wearer (at least 8 hours per day for at least 5 days per week and have had their habitual lenses no longer than 1 year). Scleral lenses wear will be defined as 15.00 mm to 19.00 mm inclusive.

Exclusion Criteria:

* Disorders that affect sensitivity (herpetic disease, severe diabetes mellitus)
* Anatomic variations of the conjunctiva that can impair proper scleral lens fitting
* Pregnancy
* Best corrected Snellen visual acuity worse than 20/30 in either eye
* Ocular pathology other than dry eye (e.g. glaucoma, macular degeneration, keratoconus) which may significantly impact visual function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Mickles, OD MS FAAO, Principal Investigator — Nova Southeastern University
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Illinois College of Optometry, Chicago, Illinois

REFERENCES:
- [Derived] Mickles CV, Harthan JS, Barnett M. Assessment of a Novel Lens Surface Treatment for Scleral Lens Wearers With Dry Eye. Eye Contact Lens. 2021 May 1;47(5):308-313. doi: 10.1097/ICL.0000000000000754. PMID 33156128

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydra-PEG Treated Lenses Followed by Untreated Lenses: Hydra-PEG treated lenses were worn for 30 days, followed a one-week washout period and then 30 days wearing untreated lenses
- Untreated Lenses Followed by Hydra-PEG Treated Lenses: Untreated lenses were worn for 30 days, followed a one-week washout period and then 30 days wearing Hydra-PEG treated lenses
Period: First Lens Type (30 Days)
Arm/Group | Hydra-PEG Treated Lenses Followed by Untreated Lenses | Untreated Lenses Followed by Hydra-PEG Treated Lenses
Started | 9 | 12
Completed | 8 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout Period (7 Days)
Arm/Group | Hydra-PEG Treated Lenses Followed by Untreated Lenses | Untreated Lenses Followed by Hydra-PEG Treated Lenses
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0
Period: Second Lens Type (30 Days)
Arm/Group | Hydra-PEG Treated Lenses Followed by Untreated Lenses | Untreated Lenses Followed by Hydra-PEG Treated Lenses
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants wore both the Hydra-PEG treated and untreated lenses in this crossover study, therefore the baseline characteristics are the same for both lens types.
Groups:
- Participants: As this was a crossover study, all participants work both the Hydra-PEG treated and untreated lenses. Therefore, the baseline characteristics were the same for both groups.
Arm/Group | Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Tear Breakup Time
Description: Tear breakup time of the ocular surface after wearing lenses
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Hydra-PEG Treated Lens Wearers: Patients wearing the Hydra-PEG treated lenses
- Untreated Lens Wearers: Patients wearing lenses without the Hydra-PEG treatment
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
seconds | 3.81 (2.63) | 2.91 (2.14)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.01, t-test, 1 sided; Paired t-test comparison

2. Primary Outcome: Corneal Fluorescein Staining
Description: Fluorescein staining followed by assessment using the Oxford grading scale (0-5, where 5 indicates the most staining and therefore the most damage to the ocular surface) of the ocular surface after wearing Hydra-PEG treated lenses compared to control lenses
Time Frame: 30 days
Population: All participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
score on a scale | 0.92 (0.79) | 1.40 (1.05)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was <0.05; Wilcoxon signed rank comparisons, one-sided

3. Primary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: Dry eye questionnaire to assess symptoms after wearing Hydra-PEG treated lenses compared to control lenses. Patients will be scored from 0 (no dry eye disease) to 100 (severe dry eye disease).
Time Frame: 30 days
Population: all participants
Measure: Mean (Standard Deviation); unit: OSDI score
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
OSDI score | 28.24 (12.90) | 35.10 (17.60)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.01, t-test, 1 sided; paired 1-sided t-test

4. Primary Outcome: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8)
Description: Validated dry eye questionnaire to assess symptoms after wearing Hydra-PEG treated lenses compared to control lenses. Scale is from 1 to 37, with higher scores indicating more dry eye symptoms.
Time Frame: 30 days
Population: all participants
Measure: Mean (Standard Deviation); unit: CLDEQ-8 score
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
CLDEQ-8 score | 11.89 (5.26) | 17.30 (6.50)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); Wilcoxon signed rank comparison, one sided p value

5. Secondary Outcome: Tear Breakup Time Over the Surface of the Scleral Lens
Description: Tear breakup time over the surface of the Hydra-PEG treated scleral lens compared to the control lens
Time Frame: 30 days
Population: all participants
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
seconds | 5.88 (5.17) | 4.75 (2.82)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p > 0.05, t-test, 1 sided — Calculated p value was >0.05; paired

6. Secondary Outcome: Lid Wiper Epitheliopathy
Description: Fluorescein and lissamine staining to assess lid wiper epitheliopathy using a grading scale to see if there is a change in the height and width of the staining of the lid wiper area with Hydra-PEG treated lenses compared to untreated control lenses. The lid wiper area is the portion of the marginal conjunctival epithelium of the upper eyelid that wipes the ocular surface or lens during blinking. Epitheliopathy is scored on a scale from 0 (best patient outcome) to 3 (worst patient outcome, more staining) on the basis of the horizontal and vertical extent of lid margin staining.
Time Frame: 30 days
Population: all participants analyzed with each lens type
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
score on a scale | 0.89 (0.76) | 1.41 (0.62)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was <0.05; paired, 1-sided

7. Secondary Outcome: Contact Lens-related Papillary Conjunctivitis
Description: Visual inspection for contact lens-related papillary conjunctivitis with scoring by the Efron grading scale for papillary conjunctivitis [0 (normal) to 4 (severe)] to assess changes after wear of Hydra-PEG treated lenses compared to control lenses.
Time Frame: 30 days
Population: all participants were analyzed in each lens type
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
score on a scale | 0.89 (0.66) | 1.45 (0.51)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); paired, 1-sided

8. Secondary Outcome: Temporal Conjunctival Lissamine Green Staining
Description: Temporal conjunctival lissamine green staining scored 0 (no staining) to 4 (most staining).
Time Frame: 30 days
Population: all participants analyzed in both lens types
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
score on a scale | 0.95 (0.79) | 1.23 (1.03)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was <0.05; paired, 1-sided

9. Secondary Outcome: Nasal Conjunctival Lissamine Green Staining
Description: Nasal conjunctival lissamine green staining scored from 0 (no staining) to 4 (most staining).
Time Frame: 30 days
Population: all participants were analyzed in both lens types
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydra-PEG Treated Lens Wearers | Untreated Lens Wearers
Number analyzed (Participants) | 19 | 19
score on a scale | 0.79 (0.71) | 1.03 (0.98)
Statistical Analysis 1: Comparison: Hydra-PEG Treated Lens Wearers vs Untreated Lens Wearers; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney) — Calculated p value was >0.05; paired, 1-sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the period of the study (a period of 79 days for each participant).
Groups:
- Hydra-PEG Treated Lenses Followed by Untreated Lenses: Participants wore Hydra-PEG lenses for 30 days, followed by a 7 day washout period and then 30 days wearing untreated lenses.
- Untreated Lenses Followed by Hydra-PEG Treated Lenses: Participants wore untreated lenses for 30 days, followed by a 7 day washout period and then 30 days wearing Hydra-PEG treated lenses.
Arm/Group | Hydra-PEG Treated Lenses Followed by Untreated Lenses | Untreated Lenses Followed by Hydra-PEG Treated Lenses
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI has the right to publish results from the study. The Sponsor has 30 days to review communications prior to publication with respect to the disclosure of confidential information (study results would not qualify as confidential information).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT03417505/Prot_SAP_000.pdf